CLINICAL TRIAL: NCT06711770
Title: Characterization of the Effect of G-CSF on the Interactions Between MDSC and Cancer Stem-cells in Non-small Cell Lung Cancers (CIRCUIT)
Brief Title: Effect of G-CSF on MDSC and Cancer Stem-cells Interactions in Non-small Cell Lung Cancers (CIRCUIT)
Acronym: CIRCUIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHUBX 2023/54
Record Dates: First submitted 2024-10-09; First posted 2024-12-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer; Immunotherapy; Granulocyte Colony Stimulating Factor
Keywords: Non-small cell lung cancer; Immunotherapy; Myeloid-Derived Suppressor Cells; Granulocyte-Colony Stimulating Factor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving G-CSF (Other)
  Interventions: Biological: Blood sample
- Patients without G-CSF (Other)
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Four tubes of 7 mL collected at baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months and 24 months (end of chemo-immunotherapy) or in case of relapse

SUMMARY:
Immunotherapy have revolutionized the field of oncology, but response rates are low and all patients relapse, due to immunologic (myeloid immunosuppressive cells) and non-immunologic (cancer stem- cells (CSC)) mechanisms. CSC are able to circulate within blood, protected from destruction by immunosuppressive cells such as MDSC. Some factors such as G-CSF, administered to lower febrile neutropenia, should modulate properties of MDSC and CSC, but data are contradictory, and literature remain poor regarding its effects on the interactions between MDSC and CSC in blood clusters. Indeed, this project aims at better characterizing the effect of G-CSF on these interactions and on their functions in NSCLC patients receiving G-CSF.

DETAILED DESCRIPTION:
MDSC, CSC and the clusters in blood from NSCLC patients will be assessed to evaluate the impact of G-CSF on their phenotype and functions. Samples from 2 groups of NSCLC patients receiving chemotherapy and immunotherapy will be used: 15 receiving concomitant G-CSF, and 15 not receiving concomitant G-CSF

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) aged ≥ 18 years
* Histological or cytological proven lung adenocarcinoma, metastatic or locally advanced not accessible to local therapy
* Receiving chemotherapy and immunotherapy as first-line treatment
* Signed written informed consent (no later than the day of inclusion, and before the blood sample collection)
* Patient affiliated or beneficiary to a health security system;

Exclusion Criteria:

* Patient with a small cell lung carcinoma
* Non-metastatic disease
* Actionable mutation or genomic alteration in EGFR, ALK or ROS1
* Corticosteroids > 10 mg/j
* Autoimmune disease
* Active and uncontrolled HIV infection
* Concomitant cancer
* Pregnancy or lactating women
* Psychiatric or medical conditions that prohibit the understanding and rendering of informed consent
* Patient under a legal protection measure
* Patient with a deprived liberty condition
* Patient incapable of giving signed informed consent
* Patient within the exclusion period for another clinical trial, or participating to another interventional trial within 30 days before the beginning of this project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Phenotype of MDSC and CSC | At baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months and 24 months (end of chemo-immunotherapy) or in case of relapse
  Expression of different MDSC markers corresponding to the rate of the different MDSC subpopulations
Functions of MDSC and CSC | At baseline, 3 weeks, 6 weeks, 12 weeks, 6 months, 12 months and 24 months (end of chemo-immunotherapy) or in case of relapse
  Immunosuppressive and non immunosuppressive functions of the different populations of MDSC

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, service d'Oncologie Médicale, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No